CLINICAL TRIAL: NCT04948008
Title: A Seamless Phase IIb/III Clinical Study to Evaluate the Efficacy and Safety of IBI306 in Subjects With Homozygous Familial Hypercholesterolemia in China
Brief Title: Evaluate the Efficacy and Safety of IBI306 in Subjects With Homozygous Familial Hypercholesterolemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LQY-PCSK9-Homozygous
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Familial Hypercholesterolemia - Homozygous; Lipid Metabolism Disorders; Proprotein Convertase Subtilisin/Kexin 9
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: The first phase of this research is the randomized design of open labels. The second stage is an open, single-arm design.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1 (Experimental): The subjects received IBI306 150 mg Q2W subcutaneously injected into the abdomen each time for 12 weeks;
  Interventions: Biological: IBI306
- Treatment group 2 (Experimental): The subjects received IBI306 300 mg Q4W subcutaneously injected into the abdomen each time for 12 weeks;
  Interventions: Biological: IBI306

INTERVENTIONS:
Biological: IBI306 — IBI306 is a kind of Proprotein convertase subtilisin/kexin 9

SUMMARY:
IBI306 is a bio-innovative drug against proprotein convertase subtilisin 9 (PCSK-9) monoclonal antibody. Currently, cholesterol-lowering drugs with multiple mechanisms of action are on the market or under development. Among them, anti-PCSK-9 monoclonal antibodies have received widespread attention due to their good safety and efficacy. The results of existing preclinical studies show that IBI306 has a clear structure, good stability, and is not inferior to other drugs of its kind in terms of drug activity, animal pharmacokinetics (PK)/pharmacodynamics (PD) and safety.

This study is divided into two phases: the dose exploration phase (the first phase) and the confirmatory phase (the second phase). Each stage is divided into screening period, treatment period, and safety follow-up period. The first phase of this research is the randomized design of open labels. The second stage is an open, single-arm design.

The main purpose of the first phase of the study: to evaluate the tolerability and safety of multiple-dose repeated administration of IBI306 in the Chinese population with hypercholesterolemia, and to recommend the dose for the second phase. The main purpose of the second phase of the study: to evaluate the effectiveness of IBI306 in the Chinese homozygous familial hypercholesterolemia population. Secondary research purpose: To evaluate the safety and immunogenicity of IBI306 in Chinese homozygous familial hypercholesterolemia population.

DETAILED DESCRIPTION:
Inclusion Criteria

1. Provide a signed and dated informed consent form.
2. Men or women aged ≥18 and ≤80 at the time of screening.
3. Weight ≥40 kg at the time of screening.
4. Meet at least one of genetic testing confirmation or clinical data to diagnose homozygous familial hypercholesterolemia.

   Clinical diagnosis basis: based on untreated LDL-C concentration> 13 mmol/L or after treatment (defined as receiving moderate-strength or maximum tolerated dose of statin for at least 4 weeks, with or without ezetimibe ) LDL-C concentration> 8mmol/L, and xanthoma occurred before the age of 10 or both parents have a history of heterozygous familial hypercholesterolemia.
5. Maintain a low-fat diet and stably take the current lipid-lowering therapy (taking moderate-strength statins, except for statin intolerance, with or without ezetimibe, bile acid chelator, or niacin) for at least 4 weeks.
6. The fasting LDL cholesterol concentration of the local laboratory at the time of screening was ≥3.4 mmol/L.
7. Fasting triglycerides ≤4.5 mmol/L during screening by the local laboratory.
8. The subjects indicated their willingness and cooperation to complete all the steps in the research and the research intervention period.

Exclusion criteria

1. Dialysis or plasma exchange was performed within 8 weeks before screening.
2. Patients who have received liver transplant surgery in the past.
3. Have used Mipomethamine or Lometapide within 5 months before screening.
4. Subjects should adjust their current lipid-lowering drug regimen or doses such as statins within 4 weeks before screening (these subjects can stabilize the current dose of lipid-lowering drugs such as statins and can be re-screened for 1 month).
5. There are uncontrolled clinical diseases that may affect blood lipids or lipoprotein levels (for patients with thyroid hormone replacement therapy, the thyroid hormone dose needs to be stabilized for at least 6 weeks before the screening visit)
6. New York Heart Association (NYHA) grade III or IV heart failure, or recently detected left ventricular ejection fraction <30%.
7. Uncontrolled severe arrhythmia, defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response or supraventricular tachycardia.
8. Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting or stroke occurred within 3 months before enrollment.
9. Plan to have heart surgery or revascularization within 20 weeks after screening.
10. Poorly controlled hypertension is defined as a systolic blood pressure> 180 mmHg or a diastolic blood pressure> 110 mmHg confirmed by repeated measurements.
11. Moderate to severe renal insufficiency, defined as the estimated glomerular filtration rate <30 ml/min/1.73m2 during the screening period, calculated using the MDRD formula: eGFR =186 x SCr (mg/dl)-1.154x (age )-0.203x (0.742 [if female]), the unit conversion of blood creatinine: 1μmol/L=0.0113 mg/d.
12. Active liver disease or liver function impairment is defined as the screening period determined by local laboratory analysis, aspartate aminotransferase or alanine aminotransferase> 3 times the upper limit of normal (ULN).
13. Creatine kinase (CK) ≥ 5 times of ULN during screening, confirmed by repeated measurements at least 1 week apart.
14. As judged by the investigator, there is a known active infection or major blood, kidney, metabolic, gastrointestinal or endocrine dysfunction.
15. Diagnosed deep vein thrombosis or pulmonary embolism within 3 months before enrollment.
16. Except for those who have been sterilized or menopausal, female subjects with potential for pregnancy, if they are unwilling to inform their sexual partners to participate in the clinical study, and take effective measures during the use of the study drug and within 15 weeks after the last dose of the study drug Contraceptive measures. Male subjects are unwilling to inform their female sexual partners that they participate in the clinical study.
17. Subjects who are pregnant or breastfeeding, or planning to become pregnant or breastfeeding during the period of study medication or within 15 weeks after the last dose of study medication.
18. Suffered from malignant tumors in the past 5 years (except for non-melanoma skin cancer, cervical carcinoma in situ, ductal carcinoma in situ of the breast or stage 1 prostate cancer).
19. Human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies or syphilis antibodies were positive at the time of screening.
20. The subject has been treated with a PCSK9 inhibitor or participated in other studies that inhibit PCSK9.
21. Known allergy to study drug and its ingredients.
22. Those who are judged by the investigator to be unsuitable to participate in the study (for example, alcohol or other drug abuse, inability or unwillingness to comply with the agreement, or mental illness).
23. Currently participating in another medical device or drug research, or the previous medical device or drug clinical research has ended, but the last time to receive other research drugs is within 30 days of screening.
24. In any other circumstances, the investigator or the sponsor after discussing it may impair the subject's ability or safety to give written informed consent and/or comply with all necessary research procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form.
2. Men or women aged ≥18 and ≤80 at the time of screening.
3. Weight ≥40 kg at the time of screening.
4. Meet at least one of genetic testing confirmation or clinical data to diagnose homozygous familial hypercholesterolemia.

   Clinical diagnosis basis: based on untreated LDL-C concentration> 13 mmol/L or after treatment (defined as receiving moderate-strength or maximum tolerated dose of statin for at least 4 weeks, with or without ezetimibe ) LDL-C concentration> 8mmol/L, and xanthoma occurred before the age of 10 or both parents have a history of heterozygous familial hypercholesterolemia.
5. Maintain a low-fat diet and stably take the current lipid-lowering therapy (taking moderate-strength statins, except for statin intolerance, with or without ezetimibe, bile acid chelator, or niacin) for at least 4 weeks.
6. The fasting LDL cholesterol concentration of the local laboratory at the time of screening was ≥3.4 mmol/L.
7. Fasting triglycerides ≤4.5 mmol/L during screening by the local laboratory.
8. The subjects indicated their willingness and cooperation to complete all the steps in the research and the research intervention period.

   -

Exclusion Criteria:

1. Dialysis or plasma exchange was performed within 8 weeks before screening.
2. Patients who have received liver transplant surgery in the past.
3. Have used Mipomethamine or Lometapide within 5 months before screening.
4. Subjects should adjust their current lipid-lowering drug regimen or doses such as statins within 4 weeks before screening (these subjects can stabilize the current dose of lipid-lowering drugs such as statins and can be re-screened for 1 month).
5. There are uncontrolled clinical diseases that may affect blood lipids or lipoprotein levels (for patients with thyroid hormone replacement therapy, the thyroid hormone dose needs to be stabilized for at least 6 weeks before the screening visit)
6. New York Heart Association (NYHA) grade III or IV heart failure, or recently detected left ventricular ejection fraction <30%.
7. Uncontrolled severe arrhythmia, defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response or supraventricular tachycardia.
8. Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting or stroke occurred within 3 months before enrollment.
9. Plan to have heart surgery or revascularization within 20 weeks after screening.
10. Poorly controlled hypertension is defined as a systolic blood pressure> 180 mmHg or a diastolic blood pressure> 110 mmHg confirmed by repeated measurements.
11. Moderate to severe renal insufficiency, defined as the estimated glomerular filtration rate <30 ml/min/1.73m2 during the screening period, calculated using the MDRD formula: eGFR =186 x SCr (mg/dl)-1.154x (age )-0.203x (0.742 [if female]), the unit conversion of blood creatinine: 1μmol/L=0.0113 mg/d.
12. Active liver disease or liver function impairment is defined as the screening period determined by local laboratory analysis, aspartate aminotransferase or alanine aminotransferase> 3 times the upper limit of normal (ULN).
13. Creatine kinase (CK) ≥ 5 times of ULN during screening, confirmed by repeated measurements at least 1 week apart.
14. As judged by the investigator, there is a known active infection or major blood, kidney, metabolic, gastrointestinal or endocrine dysfunction.
15. Diagnosed deep vein thrombosis or pulmonary embolism within 3 months before enrollment.
16. Except for those who have been sterilized or menopausal, female subjects with potential for pregnancy, if they are unwilling to inform their sexual partners to participate in the clinical study, and take effective measures during the use of the study drug and within 15 weeks after the last dose of the study drug Contraceptive measures. Male subjects are unwilling to inform their female sexual partners that they participate in the clinical study.
17. Subjects who are pregnant or breastfeeding, or planning to become pregnant or breastfeeding during the period of study medication or within 15 weeks after the last dose of study medication.
18. Suffered from malignant tumors in the past 5 years (except for non-melanoma skin cancer, cervical carcinoma in situ, ductal carcinoma in situ of the breast or stage 1 prostate cancer).
19. Human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies or syphilis antibodies were positive at the time of screening.
20. The subject has been treated with a PCSK9 inhibitor or participated in other studies that inhibit PCSK9.
21. Known allergy to study drug and its ingredients.
22. Those who are judged by the investigator to be unsuitable to participate in the study (for example, alcohol or other drug abuse, inability or unwillingness to comply with the agreement, or mental illness).
23. Currently participating in another medical device or drug research, or the previous medical device or drug clinical research has ended, but the last time to receive other research drugs is within 30 days of screening.
24. In any other circumstances, the investigator or the sponsor after discussing it may impair the subject's ability or safety to give written informed consent and/or comply with all necessary research procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
LDL-C | baseline,12 weeks and 24 weeks
  Percentage decrease in LDL-C from baseline
non HDL-C | baseline,12 weeks and 24 weeks
  Percentage decrease in non HDL-C from baseline
ApoB | baseline,12 weeks and 24 weeks
  Percentage decrease in ApoB from baseline

CONTACTS AND LOCATIONS:
Overall Officials: dong shaohong, doctor, Study Chair — Shenzhen People's Hospital
Locations (1):
- xili People's Hospital, Shenzhen, Guangdong, China